CLINICAL TRIAL: NCT04151654
Title: Investigating the Effects of Footwear Suitability on Functional Performance Level and Balance in Elderly
Brief Title: Effects of Footwear Suitability on Functional Performance and Balance in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuba Maden (Other)
Responsible Party: Sponsor-Investigator, Tuba Maden, Principal Investigator, clinical research, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-06
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Aging Disorder; Aging Problems; Aging
Keywords: aged; shoe; postural balance; accidental falls

STUDY DESIGN:
Intervention Model Description: The demographic information of the individuals (age, gender, height, body weight, body mass index (BMI), educational status) were recorded. Footwear suitability was evaluated with the Footwear Assessment Score. Subjects were assessed using the Sharpened Romberg test and Single Leg Stance test for static balance, Berg Balance Scale for dynamic balance, and Timed Up and Go test for functional performance. Balance and performance tests were done with and without footwear in all individuals. The wearing duration of footwear and accompanying disease was also recorded, and crossover methods were used for assessing balance and functional tests, with and without footwear.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- assessment1 (Other): İt is assessment study. Assessment1 was evaluated for all test with and without footwear.
  Interventions: Other: Footwear Assessment Score

INTERVENTIONS:
Other: Footwear Assessment Score — It was assessed using the Sharpened Romberg test and Single Leg Stance test for static balance. It was assessed Berg Balance Scale for dynamic balance, and Timed Up and Go test for functional performance. Balance and performance tests were done with and without footwear in all individuals.

SUMMARY:
Proper footwear serves to protect the foot against external factors. Balance and functional performance are affected by the level of footwear suitability. This study was designed to investigate the effects of footwear suitability on functional performance levels and balance in the elderly.

DETAILED DESCRIPTION:
The function of proper a footwear is to protect the foot against external factors. Balance and functional performance are affected by the level of footwear suitability. Particularly in elderly who have generally balance disorders and falling, footwear suitability is very important. Thus this study was designed to investigate the effects of footwear suitability on functional performance level and balance in elderly. The Footwear Assessment Score was used to assess parameters such as the design materials for footwear (upper and base), bending point, width, height of the toe box, getting out of the foot when walking, heel height, footwear style, wearing of the heel, and the distance between the longest toe and the end of the footwear. Thus, footwear was evaluated in many parameters.

In the literature, there are studies in which footwear was evaluated in only parameter such as height of heel.

ELIGIBILITY:
Inclusion Criteria:

* Subject has not musculoskeletal injury within the last year.
* Subject has not needed gait assistance for ambulation.

Exclusion Criteria:

* History of psychiatric, neurological and cognitive diseases.
* history of visual and hearing problems.
* Has poor coordination.
* History of chronic diseases and acute pain.
* has diabetic foot.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Footwear Assessment Score | through study completion, average one hour
  It was used to assess parameters such as the design materials for footwear (upper and base), bending point, width, height of the toe box, getting out of the foot when walking, heel height, footwear style, wearing of the heel, and the distance between the longest toe and the end of the footwear. A score of 30 on the scale represents the highest suitability level and the score taken from the scale indicates the suitability level of the footwear.
Berg Balance Scale | through study completion, average one hour
  Test was used to evaluate participants' ability to maintain their balance when performing functional activities. A BERG score of 0 and 4 points for each variable assessed represents safe and independent execution of assigned tasks (normal performance), and unsafe and dependent execution of assigned tasks (unable to perform a task), respectively. This amounts to a total score of 56 points.The Turkish version of the scale was used and a cumulative score of 0-20 indicates high risk, 21-40 moderate risk and 41-56 low risk. The test was repeated twice; with and without footwear.
Functional Performance Evaluation | through study completion, average one hour
  Timed Up and Go test (TUG) was used for evaluation of the functional performance. This test is important in terms of the assessment of mobility and balance. The participants were asked to stand from a sitting position, walk 3 m, turn back and sit back to the chair again. The test shows that it is an independent and reliable, as it involves most activities in everyday life. Duration of test was recorded. the performance duration was defined as normal balance (up to 12 s), good balance (up to 10 s) impaired balance (11-20 s) impaired balance-low risk of falling (11-20 s), and high risk of falling (longer than 20 s).

SECONDARY OUTCOMES:
Sharpened Romberg | through study completion, average one hour
  Participants were asked to remain standing, on a straight line with one leg behind the other leg, leaving the arms sagging and without impairing the balance. Four measurements involving; right foot at behind with footwear, right foot at behind without footwear, left foot at behind with footwear, and left foot at behind without footwear were taken. Duration stop criteria were defined as the time it took a participant to dislocate the foot, reach the maximal duration of 30 sec, and contact the observer to avoid falling. h-Higher scores mean a better outcome.
Single Leg Stance Test | through study completion, average one hour
  Duration of standing was measured in participants standing with dangling arms, with and without footwear. Maximal duration of test is 30 sec. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: KEZBAN BAYRAMLAR, Prof. Dr., Study Director — Supervisor of Master Thesis

IPD SHARING:
Plan to Share IPD: No
The demographic information of the individuals (age, gender, height, body weight, body mass index (BMI), educational status) were recorded. The wearing duration of footwear and accompanying disease was also recorded, and crossover methods were used for assessing balance and functional tests, with and without footwear. Footwear suitability was evaluated with the Footwear Assessment Score. Subjects were assessed using the Sharpened Romberg test and Single Leg Stance test for static balance, Berg Balance Scale for dynamic balance, and Timed Up and Go test for functional performance. Balance and performance tests were done with and without footwear in all individuals.

REFERENCES:
- [Result] McPoil TG Jr. Footwear. Phys Ther. 1988 Dec;68(12):1857-65. doi: 10.1093/ptj/68.12.1857. PMID 3057521
- [Result] SIM-FOOK L, HODGSON AR. A comparison of foot forms among the non-shoe and shoe-wearing Chinese population. J Bone Joint Surg Am. 1958 Oct;40-A(5):1058-62. No abstract available. PMID 13587573
- [Result] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Result] Hatton AL, Rome K, Dixon J, Martin DJ, McKeon PO. Footwear interventions: a review of their sensorimotor and mechanical effects on balance performance and gait in older adults. J Am Podiatr Med Assoc. 2013 Nov-Dec;103(6):516-33. doi: 10.7547/1030516. PMID 24297988
- [Result] Sherrington C, Menz HB. An evaluation of footwear worn at the time of fall-related hip fracture. Age Ageing. 2003 May;32(3):310-4. doi: 10.1093/ageing/32.3.310. PMID 12720618
- [Result] Menz HB, Lord SR. The contribution of foot problems to mobility impairment and falls in community-dwelling older people. J Am Geriatr Soc. 2001 Dec;49(12):1651-6. PMID 11843999
- [Derived] Maden T, Bayramlar K, Maden C, Yakut Y. Investigating the effects of appropriate fitting footwear on functional performance level, balance and fear of falling in older adults: A comparative-observational study. Geriatr Nurs. 2021 Mar-Apr;42(2):331-335. doi: 10.1016/j.gerinurse.2021.01.001. Epub 2021 Feb 6. PMID 33561615
- See also: Monash University Physiotherapy Department — https://www.ncbi.nlm.nih.gov/pubmed/27004631
- See also: Musculoskeletal Research Centre — https://www.ncbi.nlm.nih.gov/pubmed/16424286